CLINICAL TRIAL: NCT03133871
Title: Comparison of Scanoskin With Planimetry as an Objective Measure of Vitiligo.
Brief Title: Evaluation of Scanoskin for the Assessment of Vitiligo
Status: Completed | Type: Observational
Sponsor: Chelsea and Westminster NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: C&W17/029
Record Dates: First submitted 2017-04-21; First posted 2017-04-28 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to establish whether the use of a special digital camera (SIAscopy) can provide an accurate and reliable measure of vitiligo which is at least equivalent to the current gold standard of planimetry. If so, SIAscopy could be used as an objective diagnostic and prognostic tool in the management of vitiligo patients within dermatology departments and allow a fair and accurate assessment of new potential treatments.

DETAILED DESCRIPTION:
Vitiligo is a common, disfiguring skin complaint which affects between 0.5 and 2% of the world population and which presents with de-pigmented patches of skin. Highly stigmatising it has a profound psychological impact on those affected and negatively impacts quality of life. Efficacy of current therapies which include topical steroids/calcineurin inhibitors and ultraviolet light are limited and new treatments are required. Numerous papers including the 2010 Cochrane review have highlighted the need for a consensus on outcome measures which could then facilitate meta-analyses and provide robust clinical recommendations. No standard method of measuring skin re-pigmentation has been identified to date and current best practice relies on clinician assessment and use of various non-standardised grading systems (of which there are over 40 none of which has been proven superior or accepted by the consensus of clinicians) and in addition are neither robust nor objective. Measurement of skin pigment levels can be achieved using portable devices such as Spectrophotometric Intracutaneous Analysis scope (SIAscope) using an imaging modality called ScanoskinTM. Unlike other digital methods reported in the literature, this has been validated as a quantitative measure of melanin content in the skin, it is portable, easy to use and not prohibitively expensive. The aim of this study is to determine if ScanoskinTM is equivalent to the current gold standard of planimetry (mainly used in research setting) for establishing extent of vitiligo. In addition the investigators want to assess whether it offers a more objective standardised measure of vitiligo compared with clinician assessment (current accepted best clinical practice) which could then be utilised to provide a meaningful assessment of new and existing treatment modalities. In addition the investigators will assess whether ScanoskinTM is able to identify subclinical disease which could affect clinical decisions regarding treatment strategies and also assess whether improvements in pigmentation correlate with patient satisfaction and quality of life scores.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients diagnosed with vitiligo (any form) by a Consultant Dermatologist/Specialist Dermatology trainee.
* Who undergo any form of treatment or observation.
* Informed consent for enrolment into the study.
* Referred for assessment and treatment at Chelsea & Westminster Hospital Dermatology Department.

Exclusion Criteria:

* Patients not consenting to participate.
* Patients with insufficient English to comprehend the Patient Information Sheet (regrettably we are unable to offer translation services for this scope).
* Patients without capacity to comprehend the Patient Information Sheet would be deemed unable to give informed consent and therefore not included.
* Patients unable to undertake the imaging process for whatever reason.
* Patients unable to attend for follow up assessment

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All adult patients attending outpatient dermatology clinics at Chelsea & Westminster Hospital and diagnosed with vitiligo will be invited to take part in the study
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-11-20 (Actual); Study Completion 2018-11-20 (Actual)

PRIMARY OUTCOMES:
Comparison of Scanoskin with planimetry as an objective measure of vitiligo. | 3 years
  Comparing planimetry to Scanoskin ability to work out surface area and percentage pigmentation of vitiligo lesions

SECONDARY OUTCOMES:
Determine whether Scanoskin can identify subclinical disease | 3 years
  Taking standardised Scanoskin images of unaffected skin over time to determine if Scanoskin can pick up subclinical disease
Determine whether Scanoskin can identify subclinical response to treatment | 3 years
  Comparing images to non affected areas over time

CONTACTS AND LOCATIONS:
Overall Officials: Lucy J Thomas, MBChB, Principal Investigator — Chelsea and Westminster Hospital NHS Trust; Declan Colllins, MBBS, Study Director — Chelsea and Westminster Hospital NHS Trust
Locations (1):
- Chelsea and Westminster Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes